CLINICAL TRIAL: NCT06013540
Title: Comparison Of The Efficacy Of Combination Of TAM Formula Versus Kligman Formula For Melasma At Tertiary Care Hospital,Karachi.
Brief Title: Comparison Of Efficacy Of Combination Of TAM Formula Vs Kligman Formula For Melasma.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jinnah Postgraduate Medical Centre (Other Government)
Responsible Party: Principal Investigator, Dr Khadijah Asadullah, Principal Investigator, Jinnah Postgraduate Medical Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NO.F2-81/2022-GENL/255/JPMC
Record Dates: First submitted 2023-03-22; First posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis | interventions — hydroquinone; Tretinoin; Ascorbic Acid; Fluocinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A TAM formula (hydroquinone 2%, tretinoin 0.05% and 5% vitamin C) (Experimental)
  Interventions: Combination Product: TAM formula (hydroquinone 2%, tretinoin 0.05% and 5% vitamin C)
- Group B Kligman formula (hydroquinone 4%, fluocinolone acetonide 0.01% and tretinoin 0.05%) (Experimental)
  Interventions: Combination Product: Kligman formula (hydroquinone 4%, fluocinolone acetonide 0.01% and tretinoin 0.05%)

INTERVENTIONS:
Combination Product: TAM formula (hydroquinone 2%, tretinoin 0.05% and 5% vitamin C) — TAM formula (hydroquinone 2%, tretinoin 0.05% and 5% vitamin C)
  Arms: Group A TAM formula (hydroquinone 2%, tretinoin 0.05% and 5% vitamin C)
Combination Product: Kligman formula (hydroquinone 4%, fluocinolone acetonide 0.01% and tretinoin 0.05%) — Kligman formula (hydroquinone 4%, fluocinolone acetonide 0.01% and tretinoin 0.05%)
  Arms: Group B Kligman formula (hydroquinone 4%, fluocinolone acetonide 0.01% and tretinoin 0.05%)

SUMMARY:
This study would offer the participants about the knowledge of these formula in the treatment of melasma and help the investigators in incorporating and updating the management protocols in medical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 25-65 years of age, either gender having melasma for over one month will be included in the study
* Exclusion Criteria:

  * Pregnancy, breastfeeding, taking birth control pills or plans to become pregnant during the study
  * History of cutaneous photosensitization, porphyria, and hypersensitivity to porphyrins or photodermatosis
  * History of skin pathology or condition that could interfere with the evaluation or requires the use of interfering topical or systemic therapy
  * History of uncorrected coagulation defect or is currently using anti-coagulation medication (including but not limited to heavy aspirin therapy)
  * History of sensitivity to hydroquinone or Retin-A
  * History of evidence of a compromised immune system or hepatitis

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
EFFICACY OF COMBINATION OF TAM FORMULA VERSUS KLIGMAN FORMULA IN TREATMENT OF MELASMA | Efficacy will be assesed upto 2 months.
  Efficacy will be assessed by using Modified MASI(Melasma Area and Severity Index)In MASI scoring the "area of involvement" is calculated from 0 to 6 while the intensity and homogeneity of pigmentation are scored from 0 to 4 only. (Melasma Area Severity Index)

CONTACTS AND LOCATIONS:
Locations (1):
- JPMC, Karachi, Sindh, Pakistan